CLINICAL TRIAL: NCT04056455
Title: A Phase 1 Pharmacokinetic Study of Oral Mobocertinib in Subjects With Severe Renal Impairment and Normal Renal Function
Brief Title: A Study of Mobocertinib Capsules in People With Severe Kidney Problems and People With Healthy Kidneys
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-788-1007; U1111-1236-7343 (Registry Identifier: WHO)
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Renal Impairment; Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: conditions — Renal Insufficiency | interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe Renal Impairment: Mobocertinib 80 mg (Experimental): Participants with severe renal impairment received a single dose of mobocertinib 80 mg, capsule, orally, on Day 1.
  Interventions: Drug: Mobocertinib
- Normal Renal Function: Mobocertinib 80 mg (Experimental): Participants with normal renal function received a single dose of mobocertinib 80 mg, capsule, orally, on Day 1.
  Interventions: Drug: Mobocertinib

INTERVENTIONS:
Drug: Mobocertinib — Mobocertinib capsule.
  Other Names: TAK-788; AP32788

SUMMARY:
It is hoped that mobocertinib will eventually help people with cancer with severely reduced kidney function. The main aim of this study is to learn about the levels of mobocertinib in the blood and urine of participants with severely reduced kidney function and participants with healthy kidneys. These participants do not have cancer. The information from this study will be used to work out the best dose of mobocertinib for people with cancer with severely reduced kidney function in the future.

At the first visit, the study doctor will check who can take part. Participants who can take part will be placed into 1 of 2 treatment groups. Participants with severely reduced kidney function will be in 1 group. Participants with healthy kidneys will be in the other group. Participants in both groups will receive the same treatment and the group results will be compared.

Participants from both groups will take 1 capsule of mobocertinib. They will stay in the clinic for 10 days so the study doctors can check the amount of mobocertinib in the blood and urine of these participants over time. The study doctors will also check if the participants have any side effects from this treatment.

The clinic will call the participants 30 days after they took mobocertinib to check if they have any more side effects from their treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called mobocertinib. This study is to assess the pharmacokinetic (PK) of mobocertinib and its active metabolites (AP32960 and AP32914) in participants with severe RI compared to matched-healthy participants with normal renal function.

The study will enroll approximately 24 participants. Participants will be assigned to 1 of the following 2 treatment groups:

* Severe RI: Mobocertinib 80 mg
* Normal Renal Function: Mobocertinib 80 mg

Healthy participants with normal renal function will be recruited to match severe RI by age (mean plus or minus [+-] 10 years), gender (+-2 participants per gender), and body mass index (BMI), (mean +- 10 percent [%]). All participants will be asked to take single dose of mobocertinib on Day 1.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 51 days. Participants will be contacted by telephone 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy Participants:

1. Continuous non-smoker or moderate smoker (less than or equal to [<=] 10 cigarettes/day or the equivalent) before screening. Participant must agree to consume no more than 5 cigarettes or equivalent/day from the 7 days prior to mobocertinib dosing and throughout the period of PK sample collection.
2. Body mass index (BMI) greater than or equal to (>=) 18.0 and <=39.0 kilogram per square meter (kg/m^2), at screening. Participants will be matched to RI participants by BMI (mean +- 10%) at screening. At least 50% of the participants will be required to be of BMI >=18.0 and <=35.0 kg/m^2, at screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the Investigator or designee. Has liver function tests including alanine aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline phosphatase (ALP), and total bilirubin within the upper limit of normal at screening and at check-in.
4. Baseline estimated glomerular filtration rate (eGFR) >=90 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) based on the Modification of Diet in Renal Disease (MDRD) equation at screening divided by standard body surface area (BSA) value of 1.73 m^2. For participants with non-standard BSA, the eGFR value calculated by MDRD formula will be multiplied by the individual's BSA calculated using appropriate formula and divided by 1.73 m^2.

Inclusion Criteria for Participants with RI:

1. Continuous non-smoker or moderate smoker (<=10 cigarettes/day or the equivalent) before screening. Participant must agree to consume no more than 5 cigarettes or equivalent/day from the 7 days prior to dose of mobocertinib and throughout the period of PK sample collection.
2. BMI >=18.0 and <=39.0 kg/m^2, at screening. At least 50% of the participants will be required to be of BMI >=18.0 and <=35.0 kg/m^2, at screening.
3. Aside from RI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, ECGs, and screening clinical laboratory profiles, as deemed by the Investigator or designee.
4. Baseline eGFR 15-29 milliliter (mL) not on dialysis based on the MDRD equation at screening divided by standard BSA value of 1.73 m^2. For participants with non-standard BSA, the eGFR value calculated by MDRD formula will be multiplied by the individual's BSA calculated using appropriate formula and divided by 1.73 m^2.
5. Has a diagnosis of chronic (greater than [>] 6 months), stable (no significant changes in renal function [less than [<] 30%] in the 30 days preceding screening; no acute episodes of illness within the previous 2 months due to deterioration in renal function) renal insufficiency. Participants with RI may have related medical conditions consistent with their disease (example, mild diabetes) that are stable for at least 3 months prior to screening, in the opinion of the Investigator or designee.

Exclusion Criteria

1. Positive results at screening for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
2. Positive test result for coronavirus disease 2019 (COVID-19) testing at screening or check-in.
3. Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
4. Seated blood pressure is less than 90/40 millimeters of mercury (mmHg) or greater than 180/100 mmHg at screening.
5. Healthy participants: QT interval with Fridericia's correction (QTcF) interval is >=450 millisecond (msec) in males or >=470 msec in females or has ECG findings deemed abnormal with clinical significance by the Investigator or designee at screening
6. RI participants: QTcF interval is >500 msec or has ECG findings deemed abnormal with clinical significance by the Investigator or designee at screening.
7. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements) as indicated in (Prohibitions and Concomitant Medication) for the prohibited time period.
8. Been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
9. Donation of blood or significant blood loss within 56 days prior to dosing.
10. Plasma donation within 7 days prior to dosing.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a34a

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States from 04 March 2020 to 20 April 2022.
Pre-assignment Details: Participants with severe renal impairment or normal renal function were enrolled in this study to receive a single dose of 80 mg of mobocertinib.
Period: Overall Study
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Started | 14 | 12
Safety Analysis Set (Safety Analysis Set included all participants who received the dose of study drug.) | 14 | 12
Pharmacokinetic (PK) Analysis Set (PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile.) | 13 | 12
Completed | 13 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received the dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.86) | 59.7 (3.55) | 61.7 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 12 | 26
Height [Mean (Standard Deviation); unit: cm] | 165.1 (6.53) | 171.5 (6.32) | 168.1 (7.10)
Weight [Mean (Standard Deviation); unit: kg] | 84.30 (13.712) | 88.63 (6.997) | 86.30 (11.143)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=[weight(kg)]/[height(m)^2]
  kg/m^2 | 30.896 (4.5466) | 30.108 (1.5066) | 30.532 (3.4508)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Overall number analyzed is the number of participants eligible for descriptive statistical analysis as per criteria specified in Protocol Amendment 02.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter(ng/mL)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
nanograms per milliliter(ng/mL)
  Mobocertinib | 17.1 (326) | 11.2 (69.8)
  AP32960 | 12.2 (51.4) | 7.92 (45.8)
  AP32914 | 2.24 (73.9) | 1.51 (45.4)

2. Primary Outcome: Cmax,u: Maximum Observed Unbound Plasma Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
ng/mL
  Mobocertinib | 0.188 (252) | 0.137 (106)
  AP32960 | 0.149 (53.7) | 0.0904 (63.9)
  AP32914 | 0.0112 (108) | 0.0144 (82.7)

3. Primary Outcome: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Overall number analyzed is the number of participants eligible for descriptive statistical analysis as per criteria specified in Protocol Amendment 02. Number analyzed is the number of participants with data available for analysis for the specific category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hours(hr)/mL
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 11
ng*hours(hr)/mL
  Mobocertinib: number analyzed (Participants) | 10 | 11
  Mobocertinib | 720 (97.8) | 255 (58.1)
  AP32960 | 328 (43.6) | 184 (36.7)
  AP32914: number analyzed (Participants) | 6 | 5
  AP32914 | 93.6 (73.6) | 42.3 (33.2)

4. Primary Outcome: AUCinf,u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to Infinity for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 11
ng*hr/mL
  Mobocertinib: number analyzed (Participants) | 10 | 11
  Mobocertinib | 7.61 (77.4) | 3.16 (91.9)
  AP32960 | 4.00 (53.2) | 2.15 (56.6)
  AP32914: number analyzed (Participants) | 6 | 5
  AP32914 | 0.469 (134) | 0.461 (67.3)

5. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  Mobocertinib | 463 (184) | 219 (70.3)
  AP32960 | 305 (44.4) | 159 (42.4)
  AP32914 | 43.8 (124) | 18.7 (75.0)

6. Primary Outcome: AUClast,u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  Mobocertinib | 5.10 (145) | 2.68 (105)
  AP32960 | 3.72 (53.7) | 1.82 (63.5)
  AP32914 | 0.219 (140) | 0.172 (132)

7. Primary Outcome: Combined Molar Cmax,u: Combined Molar Unbound Cmax for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
nanomolar (nM) | 0.708 (83.7) | 0.419 (85.2)

8. Primary Outcome: Combined Molar AUClast,u: Combined Molar Unbound AUClast for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar*hour(nM*hr)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
nanomolar*hour(nM*hr) | 16.9 (79.5) | 8.14 (86.2)

9. Primary Outcome: Combined Molar AUCinf,u: Combined Molar Unbound AUCinf for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*hr
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 6 | 5
nM*hr | 30.1 (49.0) | 16.8 (36.7)

10. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
hours (hr)
  Mobocertinib | 6.00 [2.00 to 96.0] | 6.00 [4.00 to 8.00]
  AP32960 | 4.00 [2.00 to 12.0] | 6.00 [2.00 to 6.00]
  AP32914 | 6.00 [2.00 to 12.0] | 6.00 [4.00 to 8.00]

11. Primary Outcome: t1/2z: Terminal Disposition Phase Half-life for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 11
hr
  Mobocertinib: number analyzed (Participants) | 10 | 11
  Mobocertinib | 28.0 (41.5) | 23.2 (24.3)
  AP32960 | 40.1 (38.7) | 31.7 (23.3)
  AP32914: number analyzed (Participants) | 6 | 5
  AP32914 | 20.6 (58.0) | 14.6 (37.8)

12. Primary Outcome: λz: Terminal Elimination Phase Rate Constant for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Description: Terminal elimination rate constant (λz) is a mathematical estimate calculated using log-linear regression of the terminal portions of a plasma concentration against time curve.
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour (1/hr)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 11
per hour (1/hr)
  Mobocertinib: number analyzed (Participants) | 10 | 11
  Mobocertinib | 0.0248 (41.5) | 0.0299 (24.3)
  AP32960 | 0.0173 (38.7) | 0.0219 (23.3)
  AP32914: number analyzed (Participants) | 6 | 5
  AP32914 | 0.0336 (58.0) | 0.0475 (37.8)

13. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Overall number analyzed is the number of participants eligible for descriptive statistical analysis as per criteria specified in Protocol Amendment 02 and for whom the terminal disposition phase could be characterized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/hr)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 10 | 11
Liters per hour (L/hr) | 111 (97.8) | 314 (58.1)

14. Primary Outcome: CLu/F: Apparent Clearance for Unbound Drug After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Overall number analyzed is the number of participants eligible for descriptive statistical analysis as per criteria specified in Protocol Amendment 02 and for whom the terminal disposition phase of total plasma mobocertinib could be characterized.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 10 | 11
L/hr | 10500 (77.4) | 25300 (91.9)

15. Primary Outcome: Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 10 | 11
Liters (L) | 4480 (85.0) | 10500 (48.4)

16. Primary Outcome: Vz,u/F: Apparent Volume of Distribution for Unbound Drug During the Terminal Disposition Phase After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 10 | 11
Liters (L) | 424000 (61.5) | 847000 (87.7)

17. Primary Outcome: CumAe: Cumulative Amount of Mobocertinib and Its Active Metabolites (AP32960 and AP32914) Excreted in the Urine
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
milligrams (mg)
  Mobocertinib | 0.271 (0.216) | 0.357 (0.200)
  AP32960 | 0.108 (0.0457) | 0.296 (0.129)
  AP32914 | 0.0360 (0.0246) | 0.0895 (0.0361)

18. Primary Outcome: Cumfe: Cumulative Fraction of Mobocertinib Excreted in the Urine
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
percentage of dose | 0.339 (0.269) | 0.446 (0.251)

19. Primary Outcome: CLR: Renal Clearance of Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 12 | 12
L/hr
  Mobocertinib | 0.694 (0.827) | 1.78 (1.57)
  AP32960 | 0.373 (0.172) | 1.77 (0.848)
  AP32914 | 0.683 (0.427) | 3.11 (1.42)

20. Secondary Outcome: Plasma Protein Binding of Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 at multiple time points (up to 24 hours) post-dose
Population: PK Analysis Set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Number analyzed is the number of participants with data available for analysis for the specific category.
Measure: Mean (Standard Deviation); unit: percentage bound
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 13 | 12
percentage bound
  Mobocertinib | 98.8 (0.287) | 98.7 (0.420)
  AP32960: number analyzed (Participants) | 12 | 12
  AP32960 | 98.7 (0.402) | 98.8 (0.401)
  AP32914: number analyzed (Participants) | 12 | 12
  AP32914 | 99.3 (0.469) | 99.2 (0.524)

21. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A Treatment-emergent Adverse Event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug up to end of study (EOS) (up to 40 days)
Population: Safety Analysis Set included all participants who received the dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
Number analyzed (Participants) | 14 | 12
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to EOS (up to 40 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Analysis Set included all participants who received the dose of study drug.
Arm/Group | Severe Renal Impairment: Mobocertinib 80 mg | Normal Renal Function: Mobocertinib 80 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/12
Other Adverse Events (participants affected / at risk) | 5/14 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impairment: Mobocertinib 80 mg (N=14) | Normal Renal Function: Mobocertinib 80 mg (N=12)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impairment: Mobocertinib 80 mg (N=14) | Normal Renal Function: Mobocertinib 80 mg (N=12)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04056455/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04056455/SAP_001.pdf